CLINICAL TRIAL: NCT03894202
Title: Assessment of the Impact of Ultra-Early Aneurysm Treatment on Outcomes in Patients With Poor Neurological Status After Intracranial Aneurysm Rupture
Brief Title: Impact of Ultra-Early Intracranial Aneurysm Treatment in SAH
Acronym: UEAT
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, George KC Wong, Clinical Professor, Chinese University of Hong Kong
Other Study IDs: GWHMRF2018001; 06170516 (Other Grant/Funding Number: Food and Health Bureau, Hong Kong)
Record Dates: First submitted 2019-03-25; First posted 2019-03-28 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ultra-early aneurysm treatment: Ultra-early aneurysm treatment is defined as definitive cerebral aneurysm treatment such as coiling or clipping within the initial twenty-four hours.
- Non-ultra-early aneurysm treatment: Non-ultra-early aneurysm treatment is defined as definitive cerebral aneurysm treatment such as coiling or clipping after the initial twenty-four hours.

SUMMARY:
This is the first prospective study in Hong Kong that recruit patients with poor neurological status after intracranial aneurysm rupture in all seven public neurosurgical services in Hong Kong. This study assesses whether ultra-early aneurysm treatment improves outcomes in patients with poor neurological status after intracranial aneurysm rupture in Hong Kong. These data are essential to understand the impact of the disease and for future service development in Hong Kong.

DETAILED DESCRIPTION:
Objectives:

1. To evaluate outcomes in patients admitted with poor neurological status after intracranial aneurysm rupture in Hong Kong;
2. To evaluate whether ultra-early aneurysm treatment improves outcomes in patients admitted with poor neurological status after intracranial aneurysm rupture.

Hypothesis to be tested: Ultra-early aneurysm treatment increases chance of favorable outcomes in in patients admitted with poor neurological status after intracranial aneurysm rupture.

Design and subjects: Prospective observational study to recruit consecutive poor grade aneurysmal subarachnoid hemorrhage patients in the seven public neurosurgical services in Hong Kong.

Study instruments: Modified Rankin Scale, Montreal Cognitive Assessment, Stroke-Specific Quality of Life, Short Form-36, Return to Work, and hospital resource utilization.

Groups: Ultra-early (within initial 24 hours) and non-ultra early aneurysm treatment.

Main outcome measures: Favorable outcome at six months. Data analysis and expected results: Comparisons are carried out with adjustments for age, sex, admission Glasgow Coma Scale, hypertension, and modality of aneurysm treatment with appropriate regression analyses.

ELIGIBILITY:
The inclusion criteria for this study are:

1. Adult patients (aged >18 years) with spontaneous subarachnoid hemorrhage
2. Admission into Hospital Authority neurosurgical services
3. The Glasgow Coma Scale on admission ≤12 (World Federation of Neurosurgical Societies Grade 4-5)

The exclusion criteria for this study are:

1. Patients are likely to leave Hong Kong shortly after episode
2. Patients (or next-of-kin as appropriate) refuse to participate into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intracranial aneurysm rupture (aneurysmal subarachnoid hemorrhage/SAH) admitted to seven public neurosurgical services in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale | 6 months
  Modified Rankin Scale (0-6): 0-2 favourable, 3-6 unfavourable, the minimum is 0, the maximum is 6, lower score is better

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | 1, 3, 6 months
  Montreal Cognitive Assessment (0-30): 0-25 cognitive impairment, 26-30 normal cognition, higher score is better
Stroke-Specific Quality of Life | 1, 3, 6 months
  Minimum is 1, maximum is 5, higher score is better
Short Form-36 | 1, 3, 6 months
  Minimum is 0, maximum is 100, higher score is better
Return-to-Work | 1, 3, 6 months
  Return to Work: Yes or No, Work Hours and Nature, minimum work hour is 0, maximum work hour is 168 per week, longer work hour is better
Hospital Resource Utilization | 6 months
  Hospital Costs in Hong Kong Dollars, minimum is 0, maximum is 10 million, lower cost is better

OTHER OUTCOMES:
Aneurysm ultra-early treatment modality | 6 months
  Modified Rankin Scale in subgroups of Microsurgical Treatment versus Endovascular Treatment, minimum is 0 and maximum is 6 and the lower the better
Neurological Status of Patients underwent Ultra-early Aneurysm Treatment | 6 months
  Modified Rankin Scale in subgroups with WFNS Grade IV versus Patients with WFNS Grade V, minimum is 0 and maximum is 6 and the lower the better
Time of Ultra-early Aneurysm Treatment | 6 months
  Modified Rankin Scale in subgroups with Aneurysm Treatment within 6 hours and between 6-24 hours, minimum is 0 and maximum is 6 and the lower the better

CONTACTS AND LOCATIONS:
Overall Officials: George KC Wong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Surgery, The Chinese University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No